CLINICAL TRIAL: NCT06588790
Title: Diagnostic Access to Self-Care and Health Services in Low and Middle Income Countries (DASH) - Phase II
Acronym: DASH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other); Centre for Infectious Disease Research in Zambia (Other); Human Sciences Research Council (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Paul Drain, Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00019143
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Malaria Infection; Pregnancy; HIV; Diabetes; Hypertension
Keywords: Rapid diagnostic testing; Rapid testing; Self-testing; HIV; Malaria; Pregnancy; Home-based testing; community-based testing; Community Health Worker; Blood pressure; Hypertension; Diabetes; RDT
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Malaria

STUDY DESIGN:
Intervention Model Description: A three-arm household-randomized controlled implementation trial to assess two community-based intervention strategies for rapid diagnostic screening/testing, as compared to passive standard-of-care clinic-based screening/testing. Enrolled households will be randomized 1:1:1 to either one of two intervention arms, or the standard-of-care arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Home-based rapid self-testing (Experimental): Participants randomized to the home-based testing arm will be provided with rapid diagnostic tests (RDTs) for priority conditions (malaria, HIV, pregnancy) that can be used on-demand and without prior approval, if/when indicated. In this study arm, testing will be conducted primarily by the participant. Participants will be taught to use applicable RDTs at the baseline visit and a stock of RDTs with instructions for use will be left in the household.
  Interventions: Other: Home-based rapid testing
- Community health worker (CHW)-facilitated rapid testing (Experimental): Participants who are randomized to the CHW-facilitated rapid testing arm will have access to in-home testing and information through the research team. The research team will include a CHW and/or nurse who has a supply of RDTs and can conduct RDT testing, if/when indicated. This study arm is intended to be similar to local CHW-facilitated healthcare delivery programs, which may vary by country. All testing that is conducted in this arm will be performed by the CHW (or research team).
  Interventions: Other: Community health worker rapid testing
- Standard of care (No Intervention): Households randomized to the standard of care arm will receive education on indications for testing for priority conditions. Participants will be instructed to seek screening/testing at the local clinic, if/when indicated. This study arm is intended to be similar to local routine health care delivery for those in the household, which may vary by country.

INTERVENTIONS:
Other: Home-based rapid testing — Participants will be provided with rapid diagnostic tests for HIV, pregnancy and malaria (in Kenya and Zambia only) for on-demand, at-home self testing if/when indicated.
  Arms: Home-based rapid self-testing
Other: Community health worker rapid testing — Participants will have access to rapid testing through a community health worker who will conduct rapid testing in the home or at a community-based location when indicated.
  Arms: Community health worker (CHW)-facilitated rapid testing

SUMMARY:
Our primary goal is to determine if on-demand, home-based rapid testing, or rapid testing done by a community health worker (CHW) results in people testing for diseases more frequently and getting care more quickly. These two testing approaches will be compared to how individuals would normally test if they were concerned about certain diseases.

The main questions the study aims to answer are:

* Do either of the testing approaches result in more people testing themselves for certain diseases when needed?
* Does self-testing at home or testing done by a community health worker increase the number of individuals receiving test results and getting care/treatment more quickly?
* Does at-home screening for high blood pressure and diabetes result in lower blood pressure and hemoglobin A1c levels (an indicator for diabetes)?

DETAILED DESCRIPTION:
Our long-term objective is to evaluate the best use case scenarios and implementation of community-based rapid testing to enhance testing adoption and case detection, accelerate linkage to care and treatment, and improve overall health outcomes. In this study, our primary objective is to determine if on-demand, home-based rapid diagnostic testing or community health worker (CHW)-facilitated rapid diagnostic testing may improve testing adoption and access to care for select infectious diseases and non-communicable diseases in Kenya, Zambia, and South Africa. This will be completed by conducting a randomized controlled trial to evaluate two testing strategies using RDTs, as compared to the standard of care.

The specific aims of this study are the following:

* Aim #1 (Primary) - To evaluate whether on-demand, home-based rapid diagnostic testing or community health worker (CHW)-facilitated rapid diagnostic testing improve testing adoption per event (or indication) for malaria or HIV in Kenya, Zambia, and South Africa.
* Aim #2 - To evaluate whether on-demand, home-based rapid testing or community health worker (CHW)-facilitated rapid testing improves the percentage of people or households receiving a test result, improving access to care, or accelerating time to diagnosis/treatment for malaria or HIV in Kenya, Zambia, and South Africa.
* Aim #3 - To evaluate whether household screening for hypertension and diabetes with appropriate referral for confirmatory testing and treatment may decrease the median blood pressure (hypertension) or hemoglobin A1c level (diabetes) during a 6-month observational period in Kenya, Zambia, and South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Resides in the household and has spent ≥1 night at the house in the prior four weeks
* Plans to reside in the house for duration of the study
* Willing and able to provide informed consent, assent, or parental consent (where needed)

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who self-report testing for Malaria and HIV | Over a period of 6 months.
  * Malaria: Participant self-report of testing for malaria (measured as ever tested between baseline and exit).
  * HIV: Participant self-report of testing for HIV (measured as ever tested after baseline).
  * Composite: Participant self-report of testing for malaria or HIV (measured as ever tested after baseline).

SECONDARY OUTCOMES:
Number of participants who self-report testing for Malaria and HIV when indicated | Over a period of 6 months.
  * Malaria: Self-report of malaria test for each testing indication event after baseline (presence of a fever after the baseline enrollment visit)
  * HIV: Self-report of HIV test for each testing indication event after baseline (possible HIV exposure as defined by screening indication)
  * Composite: Proportion of testing indication events after baseline that received appropriate screening/testing for malaria and HIV.
Time from testing to treatment initiation or linkage to care among participants who tested positive for malaria or HIV | Over a period of 6 months
  Time from testing to treatment initiation or linkage to care if/when indicated, for malaria and HIV, among those participants who had an indication for screening or testing.
Prevalence and incidence of positive malaria test results among participants asymptomatic and symptomatic for malaria among study populations in Zambia and Kenya | Over a period of 6 months.
Diagnostic accuracy of a research use only malaria test for asymptomatic or symptomatic infection, as compared to rt-PCR testing from dried blood spots | Over a period of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Drain, MD, MPH, Principal Investigator — University of Washington
Locations (3):
- Kenya Medical Research Institute, Kisumu, Kenya
- Human Sciences Research Council, Durban, South Africa
- Center for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided